CLINICAL TRIAL: NCT05565586
Title: Impact of High Dietary Fiber on Microbiome and Vaccine Responses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0450; NCI-2022-07926 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2022-09-19; First posted 2022-10-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Influenza
Keywords: Microbiome; Flu; Fiber; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High-Fiber Diet (HFD) Intervention (Experimental): Participants are expected to eat only the study meals and snacks provided
  Interventions: Dietary Supplement: High-Fiber Diet (HFD)
- Prebiotic Food-Enriched Diet (PreFED) Intervention (Experimental): Participants are expected to incorporate study snacks and meal components provided into your usual diet.
  Interventions: Dietary Supplement: Prebiotic Food-Enriched Diet (PreFED)

INTERVENTIONS:
Dietary Supplement: High-Fiber Diet (HFD) — Participants are assigned to the high fiber diet, all meals and snacks will be provided to participants during the study. This diet includes fruits, vegetables and whole grains, a maximum of 18 oz. cooked red meat (including beef, pork, and lamb) per week, and little or no processed meats or added sugars.
  Arms: High-Fiber Diet (HFD) Intervention
Dietary Supplement: Prebiotic Food-Enriched Diet (PreFED) — Participants are assigned to the prebiotic food enriched diet, participants will receive 2 prepared snacks and 1 meal component (a key prebiotic ingredient to incorporate into meals and simple recipes) each day. Participants will also receive a handout that includes key prebiotic foods to incorporate into your own diet.
  Arms: Prebiotic Food-Enriched Diet (PreFED) Intervention

SUMMARY:
To learn if diet can enhance the microbes (such as bacteria and viruses) found in your gut and improve the body's immune response to the influenza (flu) vaccine.

DETAILED DESCRIPTION:
Primary Objectives:

--To determine the feasibility of two dietary intervention strategies focused on fiber-rich and prebiotic foods prior to seasonal influenza vaccination. Feasibility is defined as ≥ 80% of subjects being compliant with the intervention.

Secondary Objectives:

* To evaluate the effects of each dietary intervention on the composition, diversity and function of the gut microbiome.
* To assess the effects of each dietary intervention on response to influenza vaccination as measured by vaccine-specific immune response.
* To assess the effects of each dietary intervention on systemic immunity.

Exploratory Objectives:

* To interrogate the overlap between the identified gut microbial and dietary patterns associated with vaccine response and those associated with excellent or poor responses to cancer immunotherapy (from our own published work and internal cohorts).
* To identify components and determinants of the gut microbiome that could be modulated to enhance vaccine response.
* To determine how modulation of the gut microbiome can be achieved through fiber and prebiotic-focused dietary changes.

ELIGIBILITY:
Inclusion Criteria:

1. MD Anderson employees with existing MRNs
2. Body Mass Index (BMI) 18.5-40 kg/m2
3. Age 18 or older
4. Intends to receive the seasonal influenza vaccine at MD Anderson through Employee Health (starting Fall of 2022)
5. Willing to adhere to the provided dietary interventions
6. Willing to provide blood and stool specimens, complete diet questionnaires and logs, and pick up food on-site within the study schedule
7. English-speaking
8. Has easy access to a scale at home, work, or in their community

Exclusion Criteria:

1. Contraindication to the recommended annual influenza vaccine
2. Medical contraindications to the intervention diet
3. Major dietary restrictions (including vegetarian or vegan diets) or food allergies
4. Unable or unwilling to undergo study procedures
5. Has diabetes mellitus requiring medical treatment
6. Has inflammatory bowel disease
7. Has a history of bariatric surgery
8. Has a history of major gastrointestinal surgery (not including appendectomy or cholecystectomy)
9. Antibiotic use within 30 days of study initiation or planned antibiotic treatment during study course
10. Habitual consumption of a high fiber diet
11. Use of a supplement containing fiber/prebiotics/probiotics within 30 days of study initiation
12. Women who are pregnant, planning to become pregnant, or who are lactating may not be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of dietary intervention prior to seasonal influenza vaccination defined as ≥ 80% of subjects being compliant with the intervention in the cohort | through study completion an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Wargo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org